CLINICAL TRIAL: NCT00149942
Title: Conversion Trial From Mycophenolate Mofetil (MMF) to Enteric-Coated Mycophenolate Sodium (EC-MPS) in Stable Transplanted Patients Suffering From GI Adverse Events While on Mycophenolate Mofetil Therapy
Brief Title: Conversion Trial From Mycophenolate Mofetil (MMF) to Enteric-coated Mycophenolate Sodium (EC-MPS) in Stable Transplanted Patients Suffering From Gastrointestinal (GI) Adverse Events While on Mycophenolate Mofetil Therapy (MMF) Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ABE01
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation; Liver Transplantation
Keywords: Enteric coated mycophenolate sodium; transplantation; gastrointestinal adverse events; Kidney and liver transplantation patients experiencing GI AEs with current MMF treatment

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

SUMMARY:
This open, single arm, explorative study aims to investigate the evolution of gastrointestinal adverse events after switch from MMF to EC-MPS in organ transplanted patients suffering from gastrointestinal adverse events while on MMF therapy.

ELIGIBILITY:
Inclusion Criteria:

* Kidney or liver transplanted patients
* Currently under MMF therapy and currently suffering from upper or lower gastro-intestinal adverse events

Exclusion Criteria:

* Recent graft rejection before the study
* Other pre-existing conditions that may cause gastro-intestinal complaints
* Use of other drugs known to cause gastro-intestinal complaints

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal adverse events before switch versus 3 months after switch

SECONDARY OUTCOMES:
Time to the first biopsy-proven rejection after conversion.
Severity of biopsy-proven rejections after conversion.
Proportion of patients who had graft loss after conversion.
Frequency of adverse events
Frequency of infections

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland